CLINICAL TRIAL: NCT06214338
Title: Blood Bioavailability of Two Different Doses of a β-alanine Supplement
Brief Title: Blood Bioavailability of Two Different Doses of a β-alanine Supplement (BIo-β)
Acronym: Bio-β
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: UCAMCFE-00035
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2023-12

CONDITIONS: Bioavailability
Keywords: β-alanine
MeSH Terms: interventions — Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dose (Experimental): 10 mg of β-alanine
  Interventions: Dietary Supplement: Low dose
- High Dose (Experimental): 20 mg of β-alanine
  Interventions: Dietary Supplement: High dose

INTERVENTIONS:
Dietary Supplement: Low dose — Consumption of a β-alanine sustained-release supplement, 10 mg by 4 intakes of 2.5, separated by 1 hour and 15 min.
  Arms: Low Dose
Dietary Supplement: High dose — Consumption of a β-alanine sustained-release supplement, 10 mg by 4 intakes of 5 separated by 1 hour and 15 min.
  Arms: High Dose

SUMMARY:
The purpose of this study is to To study the blood bioavailability of a sustained-release β-alanine granulated supplement of two different doses (10 g and 20 g).

DETAILED DESCRIPTION:
Subjects will consume 10 g of β-alanine one day by 4 ingestions of 2.5 g separated by 1 hour and 15 min. While on another day 20 g of β-alanine by 4 ingestions of 5 g separated by 1 hour and 15 minutes, with a washout period of 15 days between the two doses. Subsequently, the amino acid levels in blood will be analyzed after the product intake and during a period of 8 hours.

Each day of visit the paresthesias (moment of appearance, intensity and sensations) will be studied at different times.

ELIGIBILITY:
Inclusion Criteria:

* Men between 18 and 60 years old.
* Cyclists with more than two years of cycling experience.
* Bicycle training at least twice a week.

Exclusion Criteria:

* Suffer a lasting injury that prevents you from training in the month prior to surgery.
* Subjects with a chronic illness.
* Having consumed in the three months prior to the start of the study any β-alanine supplement.
* Making changes in diet or exercise during the study.
* Inability to understand the informed consent form.
* Consumption of other supplements that could alter the results of the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Aminoacids in plasma | After the first intake of the product, samples will be taken at 15, 30, 45, 60 and 75 minutes. After the fourth and last product intake, samples will be taken at 15, 30, 45, 60, 75, 90, 120, 180 and 240 minutes.
  The complete series of amino acids will be analyzed in plasma, after supplement intake, for 8 hours and at various times after product intakes. A bioavailability curve will be developed for each of these samples.

SECONDARY OUTCOMES:
Paresthesia | After the first intake of the product, samples will be taken at 15, 30, 45, 60 and 75 minutes. After the fourth and last product intake, samples will be taken at 15, 30, 45, 60, 75, 90, 120, 180 and 240 minutes.
  It will be recorded by means of a visual analog scale (VAS), drawn with a continuous line of 10 centimeters where the left edge determines "no unusual sensation", translated to 0 in the recording of the data; and on the right edge "more intense sensation", translated to 10.
symptomatology - qualitative question | After the first intake of the product, samples will be taken at 15, 30, 45, 60 and 75 minutes. After the fourth and last product intake, samples will be taken at 15, 30, 45, 60, 75, 90, 120, 180 and 240 minutes.
  They should answer if they have felt at any time after the ingestion of β-alanine any symptomatology such as: prickling, itching, tingling, numbness, chills and pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No